CLINICAL TRIAL: NCT06033794
Title: Applications of Near-infrared Fluorescence Imaging Guided Lymph Node Dissection and Fluorescence Angiography of Inferior Mesenteric Artery Assisted Left Colic Artery Preservation: A Prospective Randomized Controlled Study
Brief Title: Applications of Fluorescence Imaging Guided Lymph Node Dissection and Fluorescence Angiography of Inferior Mesenteric Artery Assisted Left Colic Artery Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCC-4123
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Fluorescence; Indocyanine Green; Rectal Cancer Surgery
Keywords: Left Colic Artery; Fluorescence; No. 253 lymph node; Inferior mesenteric artery; Indocyanine green

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic No. 253 lymph node dissection and preserving the LCA under fluorescence guidance. (Experimental): Preoperatively, indoycine green fluorescent dye was injected into the anus to trace the No. 253 lymph nodes, and intraoperatively, arterial branching of the mesentery was performed by intravenous injection of fluorescent dye to preserve the left colic artery.
  Interventions: Device: Fluorescence laparoscopic system
- Performing laparoscopic No. 253 lymph node dissection and preserving the LCA. (Active Comparator): Conventional laparoscopic approach for dissection of the No. 253 lymph nodes and preservation of the left colic artery.
  Interventions: Device: Fluorescence laparoscopic system

INTERVENTIONS:
Device: Fluorescence laparoscopic system — Intraoperative fluorescence imaging was performed using the DPM-ENDOCAM-03 and DPM-LIGHT-03 fluorescence imaging system (manufactured by Digital Precision Medicine Technology Co., Ltd., Zhuhai, China). This system provides original fluorescence mode, color mode, and fusion mode, allowing real-time quantitative analysis of the fluorescence signals.

SUMMARY:
To investigate the accuracy of fluorescence angiography technique IMA classification and the impact of lymph node mapping technique on the dissection of No. 253 lymph nodes.

DETAILED DESCRIPTION:
Multiple studies, including randomized controlled trials (RCTs), have demonstrated that lymph node imaging techniques can effectively increase the number of harvested lymph nodes in gastric and colorectal cancer surgeries . However, there remains a scarcity of research specifically focused on the surgical procedure of fluorescent-guided clearance of No. 253 lymph nodes. Most existing studies have been retrospective analyses, and the need for prospective studies is evident. Further clinical research is crucial to explore the successful application of fluorescence lymph node imaging combined with indocyanine green (ICG) fluorescence angiography and its multifunctional fusion. To address this gap, investigators plan to conduct a randomized controlled trial comparing the outcomes between the use of ICG Fluorescence lymph node Imaging combined with Fluorescence angiography (FIFA group) and conventional techniques (non-ICG group) in laparoscopic rectal cancer surgery. Specifically, investigators focus will be on the preservation of the left colic artery (LCA) and the clearance of No. 253 lymph nodes. The primary objectives of our study are to simplify surgical procedures, enhance surgical safety, and provide substantial evidence for the further promotion and adoption of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Colonoscopic biopsy confirmed colorectal adenocarcinoma
* The tumor was located in the rectum or upper rectum, and the surgical method was Dxion
* No local complications before operation (no obstruction, incomplete obstruction, no massive active bleeding, no perforation, abscess formation, no local invasion)
* Preoperative imaging diagnosis was cT1-4aNxM0
* The hematopoietic functions of heart, lung, liver, kidney and bone marrow meet the requirements of surgery and anesthesia
* Sign the informed consent form

Exclusion Criteria:

* Previous surgical history of malignant colorectal tumors
* The surgical methods were combined abdominoperineal resection, Hartman operation and ISR operation
* There are contraindication of laparoscopic surgery, such as severe cardiopulmonary insufficiency
* Patients who have undergone multiple abdominal and pelvic surgeries or extensive abdominal adhesion
* Patients with intestinal obstruction, intestinal perforation, intestinal bleeding and other emergency operations
* ASA grade ≥IV and/or ECOG physical status score ≥2 points
* Patients with severe liver and kidney function, cardiopulmonary function, coagulation dysfunction or combined with serious underlying diseases can not tolerate surgery
* Have a history of serious mental illness
* Patients with uncontrolled infection before operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
success rate of IMA fluorescence imaging | From the beginning to the end of the surgery.
  ICG solution was prepared at a concentration of 2.5 g/L. A dose of 0.05 mg-0.10 mg/kg body weight of ICG was administered intravenously through a peripheral or central vein. Before the injection of ICG, the fluorescence laparoscope was set to the original fluorescence mode to monitor the IMA region in real-time.Record the success or failure rate of IMA fluorescence imaging in the observation group. Classify the successful IMA fluorescence imaging results into four different types according to the Morro classification and calculate the proportion of each type in successful imaging.

SECONDARY OUTCOMES:
Left colic artery retention rate | From the beginning to the end of the surgery.
  Recording whether the left colic artery is preserved during surger.
Incidence of IMA bleeding events | From the beginning to the end of the surgery.
  Document incidents of mesenteric artery or vein bleeding caused by vascular injury during surgery.
No.253 lymph node dissection time | From the beginning to the end of the surgery.
  Measured based on surgical videos.
Operation time | From the beginning to the end of the surgery.
  Data obtained from anesthesia records.
Intraoperative blood loss | From the beginning to the end of the surgery.
  Data obtained from anesthesia records.
Protective ostomy rate | From the beginning to the end of the surgery.
  Data obtained from surgical records.
Complication rate within 30 days after operation | within 30 days after operation.
  According to the Clavien-Dindo classification system, complications were categorized into five grades. The postoperative status of each patient was recorded within 30 days, and the proportion of complications in each grade was calculated as a percentage of the total number of observations.
Assessment of postoperative anal function urinary function within 30 days | Assessment conducted once before surgery, on postoperative day 7, and on postoperative day 30.
  Evaluation of Low Anterior Resection Syndrome (LARS) scale, assessed using the following scales at preoperative, postoperative day 7, and day 30. Scores range from 0 to 42, with lower scores indicating better outcomes.
Measurement of residual urine volume in the bladder. | On the day the catheter was removed after surgery.
  Bladder residual urine volume was measured on the same day as catheter removal. A bladder residual urine volume of less than 50 ml was considered indicative of good bladder function, while a volume greater than or equal to 50 ml was considered indicative of urinary retention.
Arterial development time | From the beginning to the end of the surgery.
  Measured based on surgical videos.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China